CLINICAL TRIAL: NCT06004232
Title: Prenatal Yoga to Prevent Postpartum Depression (PRY-D)
Brief Title: Prenatal Yoga to Prevent Postpartum Depression
Acronym: PRY-D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Amy Loree, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH131573 (NIH); R34MH131573 (NIH)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Depression
Keywords: Postpartum; Depression; Prenatal; Pregnant; Yoga; Mindfulness; Embodiment
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Methods; Therapeutics

STUDY DESIGN:
Intervention Model Description: PRY-D intervention vs treatment as usual (TAU)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRY-D intervention (Experimental): Participants in the intervention group will complete 8 prenatal yoga sessions (1x/week) in a virtual group format. The first session will be in person, in which they will meet the instructor, connect with one another through brief introductions, receive their yoga practice materials, practice basic yoga poses, and be given the schedule for the remaining sessions, including virtual access links (e.g., Webex).
  Interventions: Behavioral: Prenatal Yoga to Prevent Postpartum Depression (PRY-D) intervention
- Treatment as Usual (TAU) (Active Comparator): Participants in the the TAU group will receive routine prenatal care, during which time all patients are given information on the importance of physical activity during pregnancy.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Prenatal Yoga to Prevent Postpartum Depression (PRY-D) intervention — The PRY-D curriculum is a mindfulness-based prenatal yoga intervention which utilizes techniques to build both embodiment and mindfulness, and has previously been shown to reduce depression in a small sample of pregnant women with clinical depression.
  Arms: PRY-D intervention
Behavioral: Treatment as Usual (TAU) — TAU involves routine prenatal care, during which time all patients are given information on the importance of physical activity during pregnancy.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Although psychological interventions exist for the prevention of PPD, a yoga-based intervention to prevent PPD among at-risk women utilizes a similar theoretical foundation (i.e., mindfulness), may be more acceptable to women of minority status, and may confer additional physical activity benefits. The purpose of this pilot study is to determine the effectiveness of using a virtually delivered prenatal yoga intervention for the prevention of PPD among at-risk women in a diverse health care system and explore preliminary factors which influence implementation of the intervention. This study has 2 phases: Phase 1 will evaluate facilitators and barriers to intervention implementation among patient, clinician, and health system stakeholders, followed by an open trial, and Phase 2 will include conducting an 8-session pilot randomized controlled trial to assess the feasibility and acceptability of the proposed prenatal yoga intervention among women with a history of depression, as well as the onset and course of PPD and mediating factors. The specific aims are to: 1) Optimize delivery of a yoga intervention within a healthcare system to prevent PPD through examining facilitators and barriers of implementation, 2) Examine feasibility, acceptability and satisfaction of the intervention within a health care system, and 3) Evaluate preliminary effectiveness of the intervention on PPD and proposed mechanisms. For Phase 1, separate focus groups with patient stakeholders and clinician and administrative stakeholders will inform intervention implementation, and an open trial to refine and optimize the intervention. For Phase 2, women with a history of depression who are 8-28 weeks pregnant will be randomized to the intervention group (n=24) or treatment-as-usual (n=24) and will complete survey measures at baseline, post-intervention, and 1 and 3 months postpartum. It is hypothesized that the intervention will be feasible and acceptable, engage women of racial/ethnic minority status, and contribute to lower rates of PPD onset. Embodiment and mindfulness are the proposed mediators. Knowledge gained from this study can support prevention efforts for PPD and improve the adverse public health impact of this disorder.

DETAILED DESCRIPTION:
Postpartum depression (PPD) affects approximately 13% of women, contributing to poorer overall maternal psychological health, as well as adverse infant health, behavior, and emotional development. Women with a history of depression are 21 times more likely to experience PPD, which most commonly occurs within 4 weeks of delivery. Intervening in pregnancy to prevent the onset of perinatal mental health disorders can ameliorate these adverse outcomes and contribute to significant cost savings at $32,300/affected woman. Despite evidence-based prenatal preventive mental health services for depression, there are barriers to access, and these services do not offer the adjunctive benefits provided by yoga-based interventions, including shorter labor duration and increased likelihood of vaginal birth. Yoga interventions during pregnancy have been shown to significantly improve depressive symptoms in pregnancy. Yet, previous work examining prenatal yoga was not prevention-focused; prior studies of prenatal yoga for depression have only examined treatment for women with current depression or did not evaluate PPD. Because nearly half of women with a history of depression who develop PPD did not exhibit depressive symptoms in pregnancy, it is important to include this high-risk group in preventive interventions.

Yoga is more beneficial than other physical activity interventions for depression symptoms, including fatigue and stress, and PPD interventions yield greater benefits with targeted populations. Specifically, yoga may prevent PPD through embodiment-facilitated improvements in body image and increasing mindfulness. Yet, there are several gaps in examining effectiveness of yoga for preventing PPD: 1) although racial/ethnic minority women have higher rates of PPD than White women, they are significantly less likely to initiate treatment for PPD; yoga interventions may be more engaging; 2) generalizability of previous studies of prenatal yoga for depression have also been limited by excluding women with particular psychiatric disorders and/or excluding women already practicing yoga. Expanding this evidence-based practice to women vulnerable to developing PPD (i.e., those with a history of depression) within a health care system may be effective for engaging high-risk women in a preventive intervention to decrease the risk of PPD. The proposed study focuses on preventing PPD and improving generalizability by delivering a virtual prenatal yoga intervention for at-risk, racially diverse women in a health care system.

The proposed study seeks to pilot test the effectiveness of an adapted evidence-based, virtually-delivered 8-session group prenatal yoga pilot preventive intervention for women at high risk of PPD (i.e., history of depression) to assess onset and evaluate factors which influence implementation within a health care system. The intervention incorporates evidence-based integrated yoga with mindfulness and embodiment techniques (i.e., proposed mechanisms). The investigators will also promote the inclusion of individuals of racial/ethnic minority status in yoga interventions by assessing strategies for inclusion of these individuals from patient stakeholders. Pregnant participants with a history of depression will be recruited from Henry Ford Health (HFH), a metropolitan health system that delivers prenatal care for diverse women (29% non-Hispanic Black). The inclusion of patient, provider, and administrative stakeholders will inform recruitment, engagement, and delivery of the intervention, facilitating scalability and sustainability by assessing barriers and facilitators to implementation.

The specific aims are to:

1. Optimize a yoga intervention to prevent PPD within a healthcare system.

1.a. Examine facilitators and barriers of implementation. Conduct 3 focus groups with patient (n=6-10 pregnant women in each group with a history of depression) and qualitative interviews administrative (n=10-15 HFH women's health clinicians and administrators) stakeholders to assess logistics, engagement of racially/ethnically diverse women with a history of depression, and sustainability of the intervention. Phenomenological analyses will be used to analyze qualitative findings to increase patient-centeredness.

1. b. Optimize delivery. An open trial of pregnant women (n=14) will aid in refining intervention delivery.
2. Examine feasibility, acceptability, and satisfaction of the intervention within a health care system. Pregnant women (n=48) with a history of depression will be randomized to the intervention (n=24) or treatment as usual (TAU; n=24). Feasibility will be assessed by measuring enrollment, retention across follow-up time points, and engagement (e.g., attendance at yoga sessions) rates. A post-intervention survey will measure acceptability and satisfaction. The investigators hypothesize that the intervention will be effective for engaging racial/ethnic minorities and that there will be representative enrollment rates of these groups.
3. Evaluate effectiveness of the intervention on PPD and proposed mechanisms. Participants will complete measures of depression, embodiment, and mindfulness at baseline, post-intervention, and 1 and 3 months post-delivery. The investigators anticipate that the intervention group will have lower rates of PPD (primary outcome) at each follow-up time point, higher levels of mindfulness and embodiment (i.e., proposed mediators; a path), and that these mediators will be associated with reduced likelihood of PPD (b path).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age,
* pregnant between 8-28 weeks gestation
* receiving prenatal care at Henry Ford Health
* have a history of depression
* have an internet-enabled device with video capability for the purpose of viewing virtual yoga classes

Exclusion Criteria:

* not being fluent in English since this will be required to engage in yoga classes
* physician guidance NOT to participate in exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 1-month and 3-months postpartum
  The Edinburgh Postnatal Depression Scale (EPDS) will be used to measure presence of postpartum depression (yes/no). EPDS scores range from 0 to 30; a score of 10 or above indicates the presence of current depression symptoms.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 1-month and 3-months postpartum
  The Edinburgh Postnatal Depression Scale (EPDS) will be used to measure severity of postpartum depression (continuous). EPDS scores range from 0 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Loree, PhD, Principal Investigator — Henry Ford Health; Sara Santarossa, PhD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data from this study will be transferred to a de-identified dataset that will be available for noncommercial research use by outside investigators via a data-sharing agreement and under the auspices of the investigators. The study team will be available for support. Information related to errors in the data, future releases, and publication lists will also be shared with users.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available within 1 year after the main trial paper is published, and will be available for a period of 5 years.
Access Criteria: The data sharing agreement will include (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; (3) a commitment to destroying or returning the data after analyses are completed; and (4) a brief written plan for how the data will be used. Furthermore, users must agree to the conditions of use governing access to the data, including reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource.

REFERENCES:
- [Derived] Loree AM, Santarossa S, Coyne P, Haley EN, Boulay M, Pappas C, Braciszewski JM, Miller-Matero LR, Hicks LM. Virtually-delivered prenatal yoga to prevent postpartum depression (PRYD) in women with a history of depression: Protocol for an exploratory pilot randomized controlled trial. Contemp Clin Trials. 2025 Sep;156:108032. doi: 10.1016/j.cct.2025.108032. Epub 2025 Jul 28. PMID 40738219